CLINICAL TRIAL: NCT00207792
Title: Randomized Trial of Filgrastim Versus Placebo Following Allogeneic Bone Marrow Transplantation
Brief Title: Trial of Filgrastim Versus Placebo Following Allogeneic Bone Marrow Transplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre National de Greffe de Moelle Osseuse (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCSF
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-09

CONDITIONS: Graft vs Host Disease
Keywords: Granulocyte colony stimulating factor
MeSH Terms: conditions — Graft vs Host Disease | interventions — Filgrastim

INTERVENTIONS:
Drug: filgrastim

SUMMARY:
The effect of haematopoietic growth factors on neutrophil recovery after allogeneic bone marrow transplantation is well recognized. Recent laboratory studies demonstrated that these cytokines may also modify T-cell and dendritic cell function, but whether the effect is strong enough to alter the risk of graft-versus-host disease (GvHD) is unclear.

The aim of this randomised study is to determine the effect of granulocyte colony-stimulating factor [G-CSF] (Neupogen; filgrastim) on the risk of acute GvHD after allogeneic bone marrow transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 16 years and < 46 years
* Geno-identical allogeneic bone marrow transplantation
* Myeloablative conditioning regimen
* Haematological malignancies and acquired aplastic anemia
* Written and informed consent

Exclusion Criteria:

* ECOG performance score > 2
* T-cell depletion
* Serum creatinine level > 133 µmol/L
* Abnormal liver function
* Positive HIV test
* Pregnant women

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Ben Othman, MD, Principal Investigator — Centre National de Greffe de Moelle Osseuse
Locations (1):
- Centre National de Greffe de Moelle Osseuse, Tunis, Tunisia